CLINICAL TRIAL: NCT06827132
Title: A Non-interventional Study Evaluating Samples From Patients With Suspected Non-small Lung Cancer or Breast Cancer to Describe Pathology Practices and to Evaluate Computational Pathology Plus Artificial Intelligence Algorithms.
Brief Title: Observational Study Evaluate Pathology Practice Use Artificial Intelligence in Patient Suspected Lung and Breast Cancer
Acronym: CASCADE
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4191R00089
Record Dates: First submitted 2025-01-28; First posted 2025-02-14 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer; Breast Cancer
Keywords: Artificial intelligence; Computational Pathology; Algorithm; Positive predictive value; Negative predictive value; Galen™ Breast application; MindPeak GmBH; Laboratories
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A multinational observational study to evaluate the current pathology practices and the utilization of computational pathology plus artificial intelligence algorithms in patients with suspected lung and breast cancer.

DETAILED DESCRIPTION:
A non-interventional study evaluating samples from patients with suspected non-small lung cancer or breast cancer to describe pathology practices and to evaluate computational pathology plus artificial intelligence algorithms in Australia, Brazil, Egypt, and Kenya. Use of digital and computational Artificial intelligence pathology in countries with low and high pathologist/population ratios is critical in developing a sustainable solution. The study has two parts, the first part will focus on breast cancer, and the second part will focus on lung cancer.

The laboratories have an active digital pathology setting and evaluate samples for cancer diagnosis. The centres of lung cancer part of the study will be selected at a later stage. The study will retrospectively evaluate samples from patients who have been preliminarily diagnosed with breast or lung cancer through clinical assessments and whose samples were evaluated only by using conventional workflow.

As part of the study, computational AI pathology algorithms will be implemented in each laboratory. Two AI pathology algorithms will be used in the breast cancer part of the study. Galen™ Breast application developed by Ibex Medical Analytics will be implemented in a laboratory in Australia. MindPeak Breast, developed by MindPeak GmbH will be implemented in laboratories in Brazil, Egypt, and Kenya. After implementing computational AI pathology algorithms, 150 samples evaluated for the primary objective from each laboratory for each cancer type will be evaluated using a conventional workflow plus an AI assisted workflow with human supervision and a conventional workflow plus an AI-assisted workflow without human supervision. These evaluations will be used to analyse secondary and exploratory objectives.

ELIGIBILITY:
Inclusion Criteria:Sample from adult patients (≥ 18 years) with suspected non-small cell lung cancer or invasive breast cancer or ductal carcinoma in situ.

-

Exclusion Criteria:

* Samples with the inadequate technical quality of slides (pre-analytics quality) or images, e.g., broken slides, large out-of-focus areas, slides with fixation artefacts.

  * Samples from cases that were included in the training or technical validation.
  * Sample taken by fine needle aspiration.
  * Sample sent for cytological evaluation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data from samples that meet the following inclusion criterion will be analyzed.
  • Sample from adult patients (≥ 18 years) with suspected non-small cell lung cancer or invasive breast cancer or ductal carcinoma in situ.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
primary objective | 2 years
  The duration between the biopsy-taken date/time and the biopsy-based pathological diagnosis date/time will be calculated based on the laboratory records retrospectively.
Primary Objective | 2 years
  Reading time to assess section slides for pathological diagnosis will also be extracted from the laboratory records, if relevant information was kept in the records.
exploratory objective | 2 years
  the total cost and fees related to training, for implementing digital pathology and computational AI pathology algorithms will be assessed as an endpoint.

SECONDARY OUTCOMES:
secondary objectives | 2 years
  agreement rate :PPV and NPV for computational AI pathology algorithms (with and without human supervision) when the conventional pathology workflow is the reference will also be evaluated.
exploratory objective | 2 years
  the total cost and fees related to employees for implementing digital pathology and computational AI pathology algorithms will be assessed as an endpoint.

OTHER OUTCOMES:
Secondary Objective | 2 years
  sensitivity:PPV and NPV for computational AI pathology algorithms (with and without human supervision) when the conventional pathology workflow is the reference will also be evaluated.
Secondary Objective | 2 years
  specificity: PPV and NPV for computational AI pathology algorithms (with and without human supervision) when the conventional pathology workflow is the reference will also be evaluated.
exploratory objective | 2 years
  The total cost and fees related to hardware for implementing digital pathology and computational AI pathology algorithms will be assessed as an endpoint.
Exploratory objective | 2 years
  the total cost and fees related to software for implementing digital pathology and computational AI pathology algorithms will be assessed as an endpoint.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/